CLINICAL TRIAL: NCT01025986
Title: Uveitis in Relation to Perceived Stress: A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: C. Michael Samson, MD, Principal Investigator, The New York Eye & Ear Infirmary
Other Study IDs: NYEE120309
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Noninfectious Uveitis

SUMMARY:
The purpose of this study is to conduct a prospective analysis to determine the relationship between disease activity of noninfectious uveitis and stress.

DETAILED DESCRIPTION:
Patients presenting at The New York Eye and Ear Infirmary (NYEEI) who meet the inclusion criteria will be recruited prospectively. Patients diagnosed with non-infectious uveitis will be asked to self-administer the Perceived Stress Scale (PSS) - 10, following informed consent. Patient demographics will also be collected. The presence of inflammation will be then be assessed by the investigator. Patients will be asked to complete the PSS-10 again at all subsequent standard-of-care visits within a 6-month timeframe. PSS-10 scores are obtained by reversing the scores on the four positive items (4, 5, 7 and 8), then summing across all 10 items. Patient and the investigator will be masked to the PSS scores.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age with a diagnosis of non-infectious uveitis
* Able to self-administer the Perceived Stress Scale (PSS) - 10

Exclusion Criteria:

* Diagnosis of infectious uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the New York Eye and Ear Infirmary diagnosed with uveitis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-07

CONTACTS AND LOCATIONS:
Locations (1):
- The New York Eye and Ear Infirmary, New York, New York, United States